CLINICAL TRIAL: NCT06763809
Title: A Randomized Placebo-Controlled Study to Evaluate the Effects of a Gummy and Capsule Supplement on Symptoms of Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semaine Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20670
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: PMS; Menstrual Cramp; Mood Change
Keywords: Fatigue; Bloating; Headaches/migraines; Constipation or diarrhea
MeSH Terms: conditions — Dysmenorrhea; Fatigue; Headache; Migraine Disorders; Constipation; Diarrhea | interventions — Spectrometry, Fluorescence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PMS Capsule Group (Experimental): Participants in this arm will take the PMS capsule, which contains Vitamin D3, Magnesium, Quercetin, Curcumin, Boswellia, Milk Thistle Extract, Resveratrol, and Ashwagandha.
  Interventions: Dietary Supplement: PMS Capsule
- Capsule Placebo Group (Placebo Comparator): Participants in this arm will take a placebo capsule, containing microcrystalline cellulose and other inert ingredients.
  Interventions: Dietary Supplement: Capsule Placebo
- PMS Gummy Group (Experimental): Participants in this arm will take the PMS gummy, which contains Vitamin D3, Magnesium, Quercetin, Curcumin, Lemon Balm Extract, Milk Thistle Extract, and Resveratrol.
  Interventions: Dietary Supplement: PMS Gummy
- Gummy Placebo Group (Placebo Comparator): Participants in this arm will take a placebo gummy, containing inert ingredients such as tapioca syrup, cane sugar, and citric acid.
  Interventions: Dietary Supplement: Gummy Placebo

INTERVENTIONS:
Dietary Supplement: PMS Capsule — Participants will take 2 capsules, 4 times daily, starting at the onset of PMS symptoms and continuing until symptoms subside.
  Arms: PMS Capsule Group
Dietary Supplement: Capsule Placebo — Participants will take 2 capsules, 4 times daily, starting at the onset of PMS symptoms and continuing until symptoms subside.
  Arms: Capsule Placebo Group
Dietary Supplement: PMS Gummy — Participants will take 2 gummies, 4 times daily, starting at the onset of PMS symptoms and continuing until symptoms subside.
  Arms: PMS Gummy Group
Dietary Supplement: Gummy Placebo — Participants will take 2 gummies, 4 times daily, starting at the onset of PMS symptoms and continuing until symptoms subside.
  Arms: Gummy Placebo Group

SUMMARY:
This virtual, randomized, placebo-controlled clinical trial evaluates the effectiveness of a PMS capsule and PMS gummy in alleviating premenstrual syndrome symptoms over 12 weeks. Participants will be divided into four groups, receiving either the PMS capsule, capsule placebo, PMS gummy, or gummy placebo. Efficacy will be assessed using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female 18+ years of age.
* Must be in good health with no significant chronic conditions (such as oncological or psychiatric disorders) and a BMI under 35.
* Must experience at least five of the following symptoms during their menstrual cycle:

Menstrual pain, Menstrual cramping, Increased Irritability, Mood changes, Breast tenderness, Headaches/migraines, Bloating, Fatigue, Constipation or diarrhea, Sleep disturbances

* Must have a regular menstrual cycle with a bleed week, and must be currently tracking their menstrual cycle and able to accurately predict their bleed week.
* If using hormonal contraception, must do so for at least three months before starting the trial, and remain consistent with taking it as per healthcare provider instructions during the study.
* If using hormonal contraception, must allow for a bleed week every month.
* Must agree to avoid cannabis, CBD, ashwagandha, and supplements other than multivitamins or protein powders for 24 hours prior to the study, and during the full study duration.
* Willing to refrain from OTC pain medications or supplements to target period-related symptoms during the study period.
* Must live in the United States.

Exclusion Criteria:

* Suffers from pre-existing conditions that would prevent them from adhering to the protocol.
* Anyone currently undergoing or planning to undergo during the study period, any gynecological-related procedures.
* Anyone diagnosed with Graves disease, Hashimotos or taking any medication for their thyroid.
* Anyone who has undergone any surgeries or invasive treatments in the last six months, or is planning to during the study period.
* Anyone with any allergic reactions requiring the use of an Epi-pen.
* Anyone with known severe allergic reactions, or history of allergy or intolerance to ingredients found in over-the-counter dietary, vitamin or herbal supplements.
* Anyone with any allergies or sensitivities to any of the study product ingredients.
* Anyone with known allergies to nightshades (e.g., eggplant, tomato, bell pepper, potato).
* Unwilling to follow the study protocol.
* Anyone pregnant, breastfeeding, or trying to conceive currently or for the duration of the study.

Participants will self-report that they are not pregnant.

* Current use of an extended activity hormonal contraception (examples include Depo-Provera injection, Nexplanon implant, or hormonal intrauterine devices (IUDs)).
* Currently participating in any other clinical study or planning to at any point during this study's duration.
* Anyone who has an alcohol dependency, regularly uses cannabis, or is using illicit drugs.
* Anyone with a history of substance abuse.
* Anyone who regularly takes supplements that might reduce inflammation or is planning to at any point during the study period.
* Anyone currently taking prescription pain medication for any indication.
* Anyone who is currently taking, or planning to take during the study period, any medications, supplements or products targeted at improving Premenstrual Syndrome symptoms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Premenstrual Syndrome (PMS) Symptom Severity | From baseline to Day 5 of Cycle 2 (approximately 8 weeks after baseline)
  Evaluate the effectiveness of the PMS capsule and gummy in alleviating symptoms associated with PMS, using the validated Menstrual Symptom Questionnaire (MSQ). The MSQ assesses 24 symptoms with scores ranging from 1 (never) to 5 (always), where a higher score indicates greater symptom severity.

SECONDARY OUTCOMES:
Participant Perception of PMS Symptom Relief | From baseline to Day 5 of Cycle 2 (approximately 8 weeks after baseline)
  Assess participants' subjective perception of symptom relief provided by the PMS capsule and gummy, using a custom survey with questions related to satisfaction, effectiveness, and tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No